CLINICAL TRIAL: NCT05349539
Title: Instrumental Assessment of Motor Symptoms by Means of Wearable Sensors in Patients With Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Antonio Suppa, Principal Investigator, Neuromed IRCCS
Other Study IDs: NEUR_05
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Motor Disorders
Keywords: Parkinson's disease; Wearable sensors
MeSH Terms: conditions — Parkinson Disease; Motor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Subjects: Cohort of healthy subjects as control.
- Patients with Parkinson's disease: Cohort of patients with Parkinson's disease

SUMMARY:
The clinical management of Parkinson's disease (PD) is frequently challenged by the occurrence of motor disorders and complications, such as freezing of gait, fluctuations and the ON-OFF phenomenon, primarily manifesting at home. Therapeutic decisions are usually based on periodic neurological examinations and patients' anamnestic experience collected in an outpatient setting, thus limited by several issues, including "recall bias" and subjective, semi-quantitative and operator-dependent evaluations in non-ecological settings. In the last two decades, new wearable technologies, consisting of "wireless" sensors (e.g., inertial, electromyography), have been widely applied to quantitatively assess movements in physiological and pathological conditions, even for prolonged periods in free-living settings (i.e., long-term monitoring). The aim of this study is to evaluate motor symptoms in patients with PD, such as bradykinesia, tremor, gait disturbances and balance disorders, objectively and quantitatively through the application of wearable sensors in intra- and extra hospital settings, also during common activities of daily living, in order to obtain ecological data possibly useful in the therapeutic management of the disease.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson's disease according to current consensus criteria and confirmed by follow-up clinical evaluations;
* ability to walk independently

Exclusion Criteria:

* dementia (MMSE < 24/30);
* comorbidities affecting gait (e.g., rheumatological or orthopedic issues);
* atypical parkinsonism.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include a heterogeneous cohort of patients with Parkinson's disease, with and without typical motor complications, including fluctuations and the ON-OFF phenomenon, and with and without paroxysmal gait disorders, such as freezing of gait.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Time of OFF state of therapy during daily activity hours; | 24 hours
  Time spent with poor motor control despite optimized pharmacological therapy
Number of "Wearing Off" and "ON-OFF" phenomena | 24 hours
  Number of motor complications despite optimized pharmacological therapy
Number of "freezing of gait" episodes | 24 hours
  Number of paroxysmal gait disorders despite optimized pharmacological therapy

CONTACTS AND LOCATIONS:
Locations (1):
- IRCSS Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: Undecided